CLINICAL TRIAL: NCT00000701
Title: A Phase I Evaluation of Azidothymidine (AZT) in Children With Acquired Immune Deficiency Syndrome (AIDS) or AIDS Related Complex (ARC)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: ACTG 003; Protocol 26,541-004; Project p53; 10979 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-03 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Drug Evaluation; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Zidovudine
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Zidovudine

INTERVENTIONS:
Drug: Zidovudine

SUMMARY:
The study is designed to test the drug zidovudine (AZT) in children, including study of drug levels in various parts of the body fluids, safety of the drug, and its effect on different parts of the body.

The effects of any drug, the way a drug enters the bloodstream, the way it is used by the body, and the way the body eliminates the drug may be very different in children compared with adults. The largest group of children who have AIDS are those who are less than 2 years of age. AIDS is often first identified in infants who are about 6 months old. Studies of AZT show that it might be useful in the treatment of AIDS. Thus it is important to study the effects of the drug in children.

DETAILED DESCRIPTION:
The effects of any drug, the way a drug enters the bloodstream, the way it is used by the body, and the way the body eliminates the drug may be very different in children compared with adults. The largest group of children who have AIDS are those who are less than 2 years of age. AIDS is often first identified in infants who are about 6 months old. Studies of AZT show that it might be useful in the treatment of AIDS. Thus it is important to study the effects of the drug in children.

Patients are hospitalized for 8 weeks to receive AZT through the intravenous (IV) route at 1 of 2 doses. Patients are then discharged from hospital and take AZT by mouth for 4 more weeks.

ELIGIBILITY:
Inclusion Criteria

Concurrent Treatment:

Allowed:

* Nutritional support not exceeding 120 calories/kg/day (hyperalimentation or dietary supplements including vitamin, folate, iron supplements).

Exclusion Criteria

Co-existing Condition:

Children with the following conditions are excluded:

* Asymptomatic with T-lymphocyte deficiency.
* Asymptomatic viremic patients or those not meeting definition criteria of AIDS related complex (ARC) or AIDS.
* Clinical evidence of active infection of acute nature or active significant or clinically apparent opportunistic infection at time of entry into study.
* Hemoglobinopathy including sickle cell anemia.
* Congenital infections such as toxoplasmosis or herpes simplex virus infection in the first month after birth or cytomegalovirus infection in the first 6 months after birth.

Children with the following conditions are excluded:

* Asymptomatic with T-lymphocyte deficiency.
* Asymptomatic viremic patients or those not meeting definition criteria of AIDS related complex (ARC) or AIDS.
* Clinical evidence of active infection of acute nature or active significant or clinically apparent opportunistic infection at time of entry into study.
* Hemoglobinopathy including sickle cell anemia.
* Congenital infections such as toxoplasmosis or herpes simplex virus infection in the first month after birth or cytomegalovirus infection in the first 6 months after birth.

Prior Medication:

Excluded:

* Suramin.
* Ribavirin.
* HPA 23.
* Phosphonoformate.
* Ansamycin.
* Interleukin 2.
* Interferon.
* Excluded within 30 days of study entry:
* All cytolytic chemotherapeutic agents, immunomodulating agents including steroids and immunoglobulin preparations.
* Antivirals (acyclovir, ganciclovir).

Prior Treatment:

Excluded within 4 weeks of study entry:

* Lymphocyte transfusions for immune reconstitution.
* Excluded within 3 months of study entry:
* Bone marrow transplant.

Child who is seropositive for HIV antibody or has HIV viremia and presents with one or more of following clinical criteria and at least one of the laboratory criteria may be considered an ARC patient for purpose of study:

* Clinical criteria:
* Persistent oral candidiasis despite appropriate therapy.
* Wasting syndrome characterized by failure to thrive and malnutrition.
* Recurrent or chronic unexplained diarrhea.
* Lymphadenopathy (more than 1 cm) at 2 or more noncontiguous sites.
* Hepatomegaly with or without splenomegaly.
* Encephalopathy with loss of developmental milestones and cortical atrophy present on computed tomography (CT) examination.
* Recurrent bacterial infections (bacteremia, pneumonia, septic arthritis, meningitis).
* Cutaneous anergy as defined by lack of delayed cutaneous hypersensitivity to selected antigens.
* Laboratory criteria:
* Hypergammaglobulinemia (IgG or IgA) defined as immunoglobulin values exceeding the maximum age-adjusted level.
* Decreased number of total T-lymphocytes (2 SD from mean).
* Absolute depression in T-helper cells to less than 500/mm3.
* Depressed (equal to or more than 2 SD from normal mean) in vitro mitogen response to at least one antigen.
* One positive HIV culture within 3 months of study entry into the study or blood obtained and culture pending.
* Life expectancy greater than 6 months.
* Ambulatory and free of opportunistic infection at time of entry.
* Reliably diagnosed disease at least moderately indicative of underlying cellular immunodeficiency and no known cause of underlying cellular immunodeficiency or other reduced resistance reported to be associated with that disease.
* Disease accepted as sufficiently indicative of underlying cellular immunodeficiency by CDC. In absence of these opportunistic diseases, a histologically confirmed diagnosis of chronic lymphoid interstitial pneumonitis will be considered indicative of AIDS unless test(s) for HIV are negative.

Ages: 3 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12
Dates: Study Completion 1990-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott G, Study Chair; Wilfert C, Study Chair; Pizzo P, Study Chair
Locations (2):
- United States (2):
  - Univ of Miami School of Medicine, Miami, Florida
  - Duke Univ Med Ctr, Durham, North Carolina

REFERENCES:
- [Background] Walter EB, Weinhold KJ, Wilfert CM. Enhanced p24 antigen detection in sera from human immunodeficiency virus-infected children. Pediatr Infect Dis J. 1993 Jan;12(1):94-6. doi: 10.1097/00006454-199301000-00019. No abstract available. PMID 8417433
- [Background] McKinney RE Jr, Pizzo PA, Scott GB, Parks WP, Maha MA, Lehrman SN, Riggs M, Eddy J, Lane BA, Eppes SC, et al. Safety and tolerance of intermittent intravenous and oral zidovudine therapy in human immunodeficiency virus-infected pediatric patients. Pediatric Zidovudine Phase I Study Group. J Pediatr. 1990 Apr;116(4):640-7. doi: 10.1016/s0022-3476(05)81619-1. PMID 2181102
- [Background] Dolin R, Graham BS, Greenberg SB, Tacket CO, Belshe RB, Midthun K, Clements ML, Gorse GJ, Horgan BW, Atmar RL, et al. The safety and immunogenicity of a human immunodeficiency virus type 1 (HIV-1) recombinant gp160 candidate vaccine in humans. NIAID AIDS Vaccine Clinical Trials Network. Ann Intern Med. 1991 Jan 15;114(2):119-27. doi: 10.7326/0003-4819-114-2-119. PMID 1984386
- [Background] Mitchell C, Scott G, Hutto C, Mastrucci T, Gourley J, Owens C, Sajous M. Safety and tolerance of zidovudine in pediatric AIDS. Int Conf AIDS. 1990 Jun 20-23;6(2):200 (abstract no FB488)